CLINICAL TRIAL: NCT07286786
Title: Comparison of Analgesic Efficacy of Sacral Erector Spinae Plane Block and Caudal Epidural Block in Pediatric Patients Undergoing Hypospadias Surgery
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Sümeyye, Residents in Anesthesiology, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: CemilTasciogluDr.Kankal
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group C (caudal block): Group
  Interventions: Procedure: Caudal Block Anesthesia
- Group S (sacral ESP block): Cohort
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Caudal Block Anesthesia — Caudal block, with its simple application system, high success rate (98-100%), and ability to provide reliable analgesia, is a first-line block method for pain control compared to other options, including peripheral blocks. It provides analgesic effects in the dermatomal region between T10 and S5.
  It is indicated for chronic back care in adults and for painful infraumbilical procedures such as pediatric circulation, hypospadias repair, circumcision, inguinal hernia repair, and anal atresia surgery.
  Although it is sometimes used as the sole anesthesia method in pediatric surgery, it is generally used in conjunction with general anesthesia. Congenital or therapeutic coagulation disorders should be excluded before application. Contraindications for caudal block in children include local vascular involvement, hairline cysts, and congenital spinal anomalies.
  Groups: Group C (caudal block)
Procedure: Erector Spinae Plane Block — In this block, a local anesthetic agent is injected into the fascial plane of the superficial and deep erector spinae muscle at the distal end of the transverse process of the vertebra. The aim is to block the dorsal and ventral rami of the spinal nerves. This block occurs through four different mechanisms: direct action on nerves in the fascial plane, diffusion into the paravertebral space, systemic absorption, and perforation on nerves in nearby compartments.
  Because the erector spinae muscle extends along the vertebra, ESPB can be preferred for analgesia in the neck, chest, trunk, and lower and upper extremities. With a single-level block, the local anesthetic agent spreads approximately 3-6 vertebral levels in a cranio-caudal direction. This provides guidance on the level at which the block should be performed, depending on the surgical procedure.
  Groups: Group S (sacral ESP block)

SUMMARY:
The goal of this observational study is to learn about effects of block strategies (sacral erector spinae plane block - ESP, caudal block) on perioperative pain in pediatric patients undergoing hypospadias surgery. The main question it aims to answer is:

Is there a difference in analgesic efficacy between sacral erector spinae plane block and caudal block in pediatric patients undergoing hypospadias surgery? Eighty six pediatric patients (ages 1-7 years, ASA I-II) scheduled for hypospadias repair under general anesthesia were included in this prospective randomized study. Both blocks were performed using 0.25% bupivacaine, at doses of 0.5 mL/kg for our study. Pain was assessed using the FLACC scale at 1, 2, 4, 6, 12 and 24 hours postoperatively.

DETAILED DESCRIPTION:
Postoperative pain management in pediatric urological surgery, particularly in hypospadias repair, is essential for reducing distress, minimizing analgesic requirements, and promoting early recovery. Caudal epidural block remains the gold standard for postoperative analgesia in this patient population due to its well-established safety and efficacy. However, its limitations-such as the risk of motor block, urinary retention, and unpredictable spread of local anesthetic-have encouraged the exploration of alternative regional techniques.

The sacral erector spinae plane (ESP) block, first described for thoracic and lumbar analgesia, has recently been applied in the sacral region as a novel approach for pediatric surgeries involving the perineum and genital area. The block is technically simpler, avoids the epidural space, and carries a low risk of complications. Nevertheless, data comparing its efficacy with the traditional caudal block in hypospadias surgery remain limited.

This study aimed to compare the analgesic efficacy and safety of sacral ESP block and caudal epidural block in children undergoing hypospadias repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-7 years
* Classified as ASA physical status I-II
* Scheduled for primary hypospadias repair were enrolled

Exclusion Criteria:

* Infection at the injection site
* Coagulopathy
* Spinal anomalies
* Allergy to local anesthetics
* Parental refusal.

Ages: 1 Year to 7 Years | Sex: All
Age Groups: Child
Study Population: The study included children with ASA I-II, who will undergo hypospadias surgery under general anesthesia, between 1 and 7 years of age, who have no contraindications for block application, and whose legal guardians agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
The pain status of patients in both groups will be evaluated with the FLACC score at postoperative 1, 2, 4, 6, 12 and 24 hours. | It will be evaluated at 1, 2, 4, 6, 12 and 24 hours postoperatively.
  FLACC: Face, Leg, Activity, Cry, Consolability. The FLACC score is an observational pain assessment tool used primarily in pediatric patients who are unable to communicate verbally. It evaluates pain based on five behavioral categories: 'Face, Legs, Activity, Cry, and Consolability', each scored from 0 to 2, resulting in a total score ranging from 0 to 10. A score of 0 indicates no pain, while 1-3 reflects mild pain, 4-6 moderate pain, and 7-10 severe pain. Higher FLACC scores represent poorer pain control and greater patient discomfort, whereas lower scores suggest effective analgesia and adequate patient comfort. Elevated FLACC scores are clinically significant, as they are associated with increased stress responses, agitation, fluctuations in cardiopulmonary parameters, delayed mobilization, and prolonged recovery in pediatric patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided